CLINICAL TRIAL: NCT04036617
Title: A Randomised, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of NaQuinate in Healthy Volunteers
Brief Title: Study of NaQuinate in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Haoma Medica Limited (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: HML-1/01/001
Record Dates: First submitted 2019-07-09; First posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NaQuinate (Experimental): Initial SAD cohorts will receive 1 dose between 10-150 mg. MAD cohorts will receive 7 days dosing between 70-150 mg
  Interventions: Drug: NaQuinate
- Placebo (Experimental): Initial SAD cohorts will receive 1 placebo dose between 10-150 mg . MAD cohorts will receive 7 days placebo dosing between 70-150 mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NaQuinate — SAD cohorts will receive 1 dose between 10-150 mg. MAD cohorts will receive 7 days dosing between 70-150mg
  Arms: NaQuinate
Drug: Placebo — SAD cohorts will receive 1 dose of placebo between 10-150 mg. MAD cohorts will receive 7 days dosing of placebo between 70-150mg
  Arms: Placebo

SUMMARY:
Phase 1, randomised, double-blind, placebo-controlled study of NaQuinate in healthy subjects after single ascending oral (PO) doses and multiple ascending PO doses.

DETAILED DESCRIPTION:
This first-in-human (FIH) clinical study is a Phase 1, randomised, double-blind, placebo-controlled study to assess the safety, tolerability, and PK of NaQuinate in healthy subjects after single ascending oral (PO) doses and multiple ascending PO doses.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet the following criteria will be considered eligible to participate in the clinical study:

  1. Healthy male and female subjects (women of non-childbearing potential) between 18 and 55 years of age. Note: Women of non-childbearing potential is defined as being amenorrhoeic for >12 months with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms). However, if indicated, this should be confirmed by follicle-stimulation hormone (FSH) levels consistent with menopause (according to local laboratory ranges). Or, have been permanently sterilised (e.g. hysterectomy, bilateral salpingectomy or bilateral oophorectomy).
  2. The subject is healthy as determined by past medical history and as judged by the PI or designee.
  3. The subject voluntarily agrees to participate in this study and signs an Independent Ethics Committee (IEC)-approved informed consent prior to performing any of the Screening procedures.
  4. The subject has a BMI of 18-32 kg/m2, inclusive, at Screening.
  5. The subject has no clinically significant history of previous allergy or sensitivity to NaQuinate or any of the excipients contained within the IMP.
  6. The subject has no clinically significant abnormal serum biochemistry, haematology, coagulation and urine examination values within 28 days before the first dose of IMP.
  7. The subject has no clinically significant abnormalities in 12-lead electrocardiogram (QTcF ≤ 450 mSec and PR 120-220 mSec).
  8. Male subjects and their female spouse/partner of childbearing potential must use appropriate effective methods of contraception from the time of dosing until after the end-of-study (EOS) visit. See Section 7.5.2 for protocol-specified contraception guidance.
  9. Male subjects must not donate sperm from first dose until at least 3 months after last dose of IMP.
  10. The subject is a non-smoker, defined as a subject who has not smoked previously and/or who has discontinued smoking or the use of nicotine/nicotine-containing products (including snuff and similar products) at least 3 months before the Screening visit.
  11. The subject must be available to complete the study (including all Follow-up visits).
  12. The subject must satisfy the PI / designee about their fitness to participate in the study and agree to comply with the protocol requirements, instructions, and study related restrictions

Exclusion Criteria:

* Subjects who meet one or more of the following criteria will not be considered eligible to participate in the clinical study:

  1. Female subjects who are breastfeeding or female subjects with a positive serum pregnancy test at Screening or a positive urine pregnancy test on Day -1.
  2. Subjects who have donated blood in the 3 months prior to Screening, plasma in the 7 days prior to Screening or platelets in the 6 weeks prior to Screening.
  3. A positive urine cotinine result at Screening or on Day -1.
  4. Subjects who have used the following within 7 days of first dosing: any non-prescribed systemic or topical medication (with the exception of paracetamol to a maximum of 2 g per day), remedy or supplement, any prescribed systemic or topical medication within 14 days of first dosing.
  5. Subjects who have clinically significant abnormalities in vital signs including: Systolic BP < 90 mmHG or > 140 mmHg; Diastolic BP < 50 mmHG or > 90 mmHG; Pulse rate < 45 or > 90 beats per minute.
  6. Subjects who have a history of significant drug allergy (e.g., anaphylaxis) or any clinically significant allergic condition (excluding hay fever), as determined by the PI.
  7. Any clinically significant abnormal haematology results, as determined by the PI.
  8. Subjects who have a confirmed positive urine drugs of abuse screen at Screening or Day -1, or a confirmed positive urine alcohol test at Screening or Day -1 (N.B. a positive alcohol result may be repeated at the Investigator's discretion) or subjects who are unwilling to avoid the use of alcohol within 48 hours before any study visit and while confined to the clinical unit.
  9. Subjects who received last IMP dose in a clinical study within the following time period prior to dosing: 3 months or 5 half-lives, whichever is longer.
  10. Subjects who have had a clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of dosing, as determined by the PI.
  11. A positive serology test for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies, or antibodies to human immunodeficiency virus type 1 (HIV-1) and/or type 2 (HIV 2) at Screening.
  12. Vulnerable subjects defined as individuals whose willingness to volunteer in a clinical study may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate (e.g., persons in detention, minors and those incapable of giving consent).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2019-06-18 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
To investigate the safety by assessment of AEs, of NaQuinate in healthy volunteers | approximately 8 weeks
  safety of single and multiple doses of NaQuinate as assess by the number of participants with treatment-related adverse events evaluated by the PI for their intensity, causality and severity, including Adverse events of Special interest.
To investigate the tolerability by assessment of AEs, of NaQuinate in healthy volunteers | approximately 8 weeks
  tolerability of single and multiple doses of NaQuinate as assess by the number of participants with treatment-related adverse events evaluated by the PI for their intensity, causality and severity, including Adverse events of Special interest.

SECONDARY OUTCOMES:
to Investigate the pharmacokinetics by measurment of Cmax of exposure to NaQuinate in healthy volunteers | approximately 8 weeks
  PK parameters after single or multiple dose administration measured by Cmax of exposure to NaQuninate in healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Muna Albayaty, MBChB, Principal Investigator — Parexel
Locations (1):
- Parexel Early Phase Clinical Unit - London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No